CLINICAL TRIAL: NCT02186301
Title: TIGER 1: A Randomized, Open-Label, Phase 2/3 Study of CO-1686 or Erlotinib as First-Line Treatment of Patients With EGFR-Mutant Advanced/Metastatic NSCLC
Brief Title: TIGER-1: Safety and Efficacy Study of Rociletinib (CO-1686) or Erlotinib in Patients With EGFR-mutant/Metastatic NSCLC Who Have Not Had Any Previous EGFR Directed Therapy
Acronym: EGFR
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor discontinued development of CO-1686 for NSCLC
Sponsor: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-1686-022 (TIGER-1)
Record Dates: First submitted 2014-06-30; First posted 2014-07-10 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: cancer; metastatic; locally advanced; lung; non-small cell lung cancer; NSCLC; epidermal growth factor receptor; EGFR; T790M; CO-1686; unresectable; recurrent; EGFR-directed therapy; irreversible EGFR inhibitor; TIGER; rociletinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Neoplasm Metastasis; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erlotinib Mono-Therapy (Active Comparator)
  Interventions: Drug: Erlotinib Mono-Therapy
- Rociletinib Mono-Therapy (Experimental)
  Interventions: Drug: Rociletinib Mono-Therapy

INTERVENTIONS:
Drug: Rociletinib Mono-Therapy — Rociletinib will be administered twice daily
  Arms: Rociletinib Mono-Therapy
Drug: Erlotinib Mono-Therapy — Erlotinib will be administered once a day
  Arms: Erlotinib Mono-Therapy

SUMMARY:
The purpose of this study is to compare the safety and anti-tumor effect of rociletinib with erlotinib in patients whose tumors have specific EGFR mutations and who have not previously received any treatment for advanced/metastatic EGFR mutated NSCLC. This study is a 'Randomized' Study. This means that upon entering the study, patients will be randomly assigned to be dosed with either rociletinib twice a day or erlotinib once a day. Patients will continue to take either rociletinib or erlotinib until it is no longer beneficial.

DETAILED DESCRIPTION:
This is a randomized, Phase 2/3 study of rociletinib versus erlotinib as a first-line treatment for patients with EGFR-mutant advanced/metastatic NSCLC whose tumors have EGFR-activating mutations. The study will consist of Phase 2 and Phase 3 parts which will use the same enrollment criteria and treatment assignment principles. Patients will be randomized 1:1 to erlotinib or rociletinib. The Phase 2 part is an open-label study. In the Phase 3 part, the sponsor will be blinded to the efficacy and safety results. The study will consist of a screening phase to establish study eligibility (including tumor genotype) and document baseline measurements, a treatment phase, in which patients will receive either rociletinib BID (twice a day) or erlotinib QD (once daily) to ascertain safety and efficacy until protocol-defined disease progression, and a follow-up phase, to monitor survival status and subsequent NSCLC cancer therapy. In the Phase 2 part only, patients initially randomized to erlotinib may be eligible to participate in an optional crossover phase to receive rociletinib if they demonstrate the T790M resistance mutation after radiographic progression on erlotinib treatment among other eligibility requirements. Patients eligible for this study must have EGFR-mutated NSCLC who have not been treated with an EGFR-directed therapy.Treatment with rociletinib or erlotinib is continuous. Each 28 day period of treatment will represent one cycle, with dosing initiated on Cycle 1 Day 1 (C1 D1).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed metastatic or unresectable locally advanced/metastatic NSCLC
2. Documented evidence of a tumor with activating EGFR mutations by local testing. Patients with exon 20 insertions are not eligible with the exception of patients with documented evidence of the exon 20 insertion A763_Y764insFQEA in the EGFR gene
3. Have undergone a biopsy or surgical resection of either primary or metastatic tumor tissue within 60 days of the first day of study treatment, C1D1, and have tissue available to send to sponsor laboratories or are able to undergo a biopsy during screening and provide tissue to sponsor laboratories
4. Measureable disease according to RECIST Version 1.1
5. Life expectancy of at least 3 months
6. ECOG (Eastern Cooperative Oncology Group) performance status of 0 to 1
7. Minimum age 18 years (in certain territories, the minimum age requirement may be higher (e.g. 20 years in Japan and Taiwan)
8. Adequate hematological and biological function, confirmed by defined laboratory values
9. Written consent on an IRB/IEC-approved Informed Consent Form (ICF) prior to any study-specific evaluation

Exclusion Criteria:

1. Documented evidence of an exon 20 insertion activating mutation other than A763_Y764insFQEA in the EGFR gene
2. Prior treatment with cytotoxic chemotherapy for advanced NSCLC; neoadjuvant/adjuvant chemotherapy is permitted if at least 6 months has elapsed between the end of chemotherapy and randomization
3. Active second malignancy; i.e., patient known to have potentially fatal cancer present for which he/she may be (but not necessarily) currently receiving treatment
4. Patients with a history of malignancy that has been completely treated, and currently with no evidence of that cancer, are permitted to enroll in the trial provided all chemotherapy was completed > 6 months prior and/or bone marrow transplant > 2 years prior to first day of study treatment
5. Known pre-existing interstitial lung disease
6. Brain metastases
7. Treatment with prohibited medications less than or equal to 14 days prior to first day of study treatment
8. Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval if that treatment cannot be either discontinued or switched to a different medication prior to administration of study drug
9. Prior treatment with EGFR TKIs (e.g. erlotinib, gefitinib, neratinib, afatinib, AZD9291, or dacomitinib), rociletinib or other drugs that target mutant EGFR
10. Clinically significant abnormal 12-lead ECG, QT interval corrected using Fridericia's method (QTCF) > 450 ms
11. Inability to measure QT interval on ECG
12. Personal or family history of long QT syndrome
13. Implantable pacemaker or implantable cardioverter defibrillator
14. Resting bradycardia < 55 beats/min
15. Non-study related surgical procedures less than or equal to 7 days prior to administration of study drug. In all cases, the patient must be sufficiently recovered and stable before treatment administration.
16. Females who are pregnant or breastfeeding
17. Refusal to use adequate contraception for fertile patients (females and males) for 12 weeks after the last dose of rociletinib and 2 weeks after the last dose of erlotinib
18. Presence of any serious or unstable concomitant systemic disorder incompatible with the clinical study
19. Any other reason the investigator considers the patient should not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-11; Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (74):
- United States (54):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - East Valley Hematology and Oncology Medical Group, Inc., Burbank, California
  - City of Hope, Duarte, California
  - Compassionate Cancer Care Medical Group, Inc., Fountain Valley, California
  - St. Joseph Heritage Healthcare, Fullerton, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of Southern California, Norris Comprehensive Cancer Center, Los Angeles, California
  - Sutter Medical Group, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Sansum Clinic, Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - UCLA Medical Center, Santa Monica, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Cancer Specialists of North Florida, Fleming Island, Florida
  - Florida Cancer Specialists and Research Institute, Fort Myers, Florida
  - Advanced Medical Specialties, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Northwestern University, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Harry and Jeanette Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - Walter Reed Army Institute of Research, Bethesda, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Oncology Hematology West PC, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Regional Cancer Care Associates, LLC, East Brunswick, New Jersey
  - Regional Cancer Care Associates, Morristown, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Hollings Cancer Center, Charleston, South Carolina
  - Tennessee Oncology, PLLC, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - USC/Norris Comprehensive Cancer Center, Nashville, Tennessee
  - Texas Oncology, PA, Austin, Texas
  - Texas Oncology-Beaumont, Beaumont, Texas
  - Texas Oncology, P.A., Bedford, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - The University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology-Plano East, Plano, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - University of Washington, Seattle, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - Yakima Valley Memorial Hospital, North Star Lodge, Yakima, Washington
- Germany (5):
  - Asklepios Fachkliniken München-Gauting, Gauting, Bavaria
  - Pius Hospital Oldenburg, Oldenburg, Lower Saxony
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Katholisches Klinikum Mainz, Sankt Hildegardis-Krankenhaus, Mainz, Rhineland-Palatinate
  - Evangelische Lungenklinik Berlin, Berlin
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong, New Territories
  - Queen Mary Hospital, Hong Kong
- Ospedale Civile di Livorno, Livorno, Italy
- South Korea (7):
  - Dong-A University Hospital, Busan
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea Saint Vincent's Hospital, Suwon
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
- Taiwan (3):
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou, Taoyuan District

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 subjects recruited from 74 sites, in 7 countries and randomized (1:1) to treatment with rociletinib or erlotinib.Original protocol had rociletinib starting dose of 625mg. In global Amendment 2, starting dose reduced to 500mg. Crossover to rociletinib was permitted however, only 2 patients did so. Safety data for these 2 patients are reported.
Groups:
- Rociletinib 500mg Tablets: Starting dose of 500mg. Taken orally twice daily (continuous 28 day treatment cycle). Treatment duration until radiographically confirmed disease progression.
- Rociletinib 625mg Tablets: Starting dose of 625mg. Taken orally twice daily (continuous 28 day treatment cycle). Treatment duration until radiographically confirmed disease progression.
- Erlotinib 150mg Tablets: Starting dose of 150mg. Taken orally once daily (continuous 28 day treatment cycle). Treatment duration until radiographically confirmed disease progression.
Period: Overall Study
Arm/Group | Rociletinib 500mg Tablets | Rociletinib 625mg Tablets | Erlotinib 150mg Tablets
Started | 20 | 30 | 50
Completed | 0 (Patients who are off study for any reason.) | 0 (Patients who are off study for any reason.) | 0 (Patients who are off study for any reason.)
Not Completed | 20 | 30 | 50
Not completed — Progressive Disease | 7 | 22 | 27
Not completed — Adverse Event | 5 | 5 | 5
Not completed — Death | 1 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 3
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Study Terminated by Sponsor | 1 | 0 | 11
Not completed — Protocol Deviation | 0 | 2 | 0
Not completed — Missing | 0 | 0 | 2
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rociletinib 500mg Tablets | Rociletinib 625mg Tablets | Erlotinib 150mg Tablets | Total
Number analyzed (Participants) | 20 | 30 | 50 | 100
Age, Customized [Median (Full Range); unit: years] | 66.0 [44 to 86] | 67.0 [41 to 85] | 64 [39 to 88] | 65 [39 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 32 | 67
  Male | 3 | 12 | 18 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 6 | 9
  Not Hispanic or Latino | 19 | 27 | 43 | 89
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 9 | 15 | 25 | 49
  Black or African American | 2 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 9 | 12 | 21 | 42
  Other | 0 | 0 | 1 | 1
  Missing | 0 | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 12 | 21 | 42
  Asian | 9 | 15 | 25 | 49
  Non-White, Non-Asian | 2 | 3 | 4 | 9
Number of Previous Therapies [Median (Full Range); unit: units on a scale] | 0.0 [0.0 to 1.0] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 1.0] | 0.0 [0.0 to 2.0]
Time Since Diagnosis of NSCLC [Mean (Standard Deviation); unit: months] | 7.2 (14.12) | 5.3 (10.39) | 8.2 (21.83) | 7.1 (17.57)
History of CNS Metastases [Count of Participants; unit: Participants] | 1 | 1 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) According to RECIST Version 1.1 as Determined by Investigator Review (invPFS)
Description: To compare the antitumor efficacy of oral single-agent rociletinib with that of erlotinib as measured by progression-free survival (PFS), when administered as a first-line targeted treatment to patients with EGFR-mutated, advanced NSCLC.Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.The appearance of one or more new lesions is also considered progression.
Time Frame: Cycle 1 Day 1 to End of Treatment, up to approximately 35 months
Population: Intent-to-treat: All patients randomized.
  1 patient was not included in analysis, due to discontinuation of study shortly after randomization and prior to first dose of study drug.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rociletinib 500mg Tablets | Rociletinib 625mg Tablets | Erlotinib 150mg Tablets
Number analyzed (Participants) | 18 | 30 | 50
Days | 274 [109 to NA] — Upper Confidence Limit is not available because it cannot be calculated. | 207 [112 to 260] | 390 [282 to 499]
Statistical Analysis 1: Comparison: Rociletinib 500mg Tablets; Test type: Other; Kaplan-Meier Median = 274.0, 95% CI 2-sided [lower limit 109] (Upper Confidence Limit is not available because it cannot be calculated)
Statistical Analysis 2: Comparison: Rociletinib 625mg Tablets; Test type: Other; Kaplan-Meier Median = 207.0, 95% CI 2-sided [112.0 to 260.0]
Statistical Analysis 3: Comparison: Erlotinib 150mg Tablets; Test type: Other; Kaplan Meier Median = 390, 95% CI 2-sided [282.0 to 499.0]

2. Secondary Outcome: Confirmed Response Rate
Description: Proportion of patients with a best overall confirmed response of partial response (PR) or complete response (CR) recorded from the start of the treatment until disease progression or recurrence.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions, defined by and assessed as:
  Complete Response (CR), is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR),at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter.
  Overall Response (OR),is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment was dependent on the achievement of both measurement and confirmation criteria.
Time Frame: Cycle 1 Day 1 to End of Treatment, up to approximately 35 months.
Population: Intent-to-treat: All patients randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rociletinib 500mg Tablets | Rociletinib 625mg Tablets | Erlotinib 150mg Tablets
Number analyzed (Participants) | 20 | 30 | 50
percentage of participants | 25.0 [8.7 to 49.1] | 40.0 [22.7 to 59.4] | 78.0 [64.0 to 88.5]
Statistical Analysis 1: Comparison: Rociletinib 500mg Tablets; Test type: Other; Percentage = 25.0, 95% CI 2-sided [8.7 to 49.1]
Statistical Analysis 2: Comparison: Rociletinib 625mg Tablets; Test type: Other; Percentage = 40.0, 95% CI 2-sided [22.7 to 59.4]
Statistical Analysis 3: Comparison: Erlotinib 150mg Tablets; Test type: Other; Percentage = 78.0, 95% CI 2-sided [64.0 to 88.5]

3. Secondary Outcome: Duration of Response
Description: Duration of Response in Patients with Confirmed Response per Investigator
Time Frame: Cycle 1 Day 1 to End of Treatment, up to approximately 35 months
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rociletinib 500mg Tablets | Rociletinib 625mg Tablets | Erlotinib 150mg Tablets
Number analyzed (Participants) | 5 | 12 | 39
Days | 225 [113 to NA] — Upper Confidence Limit is not available because it cannot be calculated. | 195.5 [143.0 to 617.0] | 335.0 [282.0 to 480.0]
Statistical Analysis 1: Comparison: Rociletinib 500mg Tablets; Test type: Other; Kaplan Meier Median = 225, 95% CI 2-sided [lower limit 113] (Upper Confidence Limit is not available because it cannot be calculated.)
Statistical Analysis 2: Comparison: Rociletinib 625mg Tablets; Test type: Other; Kaplan Meier Median = 195.5, 95% CI 2-sided [143.0 to 617.0]
Statistical Analysis 3: Comparison: Erlotinib 150mg Tablets; Test type: Other; Kaplan Meier Median = 335.0, 95% CI 2-sided [282.0 to 480.0]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from the time the first dose of study drug is administered, and until 28 days after the last dose. In addition, study procedure-related AEs that occur after signing of the informed consent form and before first dose of study drug were expected to be reported. Any Serious Adverse Events or Adverse Events of Special Interest were followed until resolution or stabilization, or until patient is lost to follow-up.
Description: If a subject experiences the same preferred term (system organ class) multiple times, then the subject will be counted only once for that preferred term (system organ class).
  Treatment Arm/Groups for subjects (n=2) who crossed over to Rociletinib from Erlotinib are included.
Groups:
- Crossover From Erlotinib 150mg to Rociletinib 500mg: Patients initially randomized to erlotinib were eligible to participate in an optional crossover phase to receive CO-1686.
  Starting dose of 500mg CO-1686. Taken orally twice daily (continuous 28 day treatment cycle). Treatment duration until radiographically confirmed disease progression.
- Crossover From Erlotinib 150mg to Rociletinib 625mg: Patients initially randomized to erlotinib were eligible to participate in an optional crossover phase to receive CO-1686.
  Starting dose of 625mg. Taken orally twice daily (continuous 28 day treatment cycle). Treatment duration until radiographically confirmed disease progression.
Arm/Group | Rociletinib 500mg Tablets | Rociletinib 625mg Tablets | Erlotinib 150mg Tablets | Crossover From Erlotinib 150mg to Rociletinib 500mg | Crossover From Erlotinib 150mg to Rociletinib 625mg
All-Cause Mortality (participants affected / at risk) | 3/19 | 1/30 | 2/50 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 10/19 | 15/30 | 7/50 | 0/1 | 1/1
Other Adverse Events (participants affected / at risk) | 19/19 | 30/30 | 50/50 | 0/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rociletinib 500mg Tablets (N=19) | Rociletinib 625mg Tablets (N=30) | Erlotinib 150mg Tablets (N=50) | Crossover From Erlotinib 150mg to Rociletinib 500mg (N=1) | Crossover From Erlotinib 150mg to Rociletinib 625mg (N=1)
Diabetic ketoacidosis (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Endocrine disorders) | 1 | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Torsade de pointes (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Acute cholangtis, Acute cholecystitis and acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Catheter site haematoma (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 2 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rociletinib 500mg Tablets (N=19) | Rociletinib 625mg Tablets (N=30) | Erlotinib 150mg Tablets (N=50) | Crossover From Erlotinib 150mg to Rociletinib 500mg (N=1) | Crossover From Erlotinib 150mg to Rociletinib 625mg (N=1)
Combined Terms of Hyperglycemia (Endocrine disorders) | 10 | 16 | 3 | 0 | 0
Combined Terms of QTc Prolongation (Cardiac disorders) | 2 | 8 | 1 | 0 | 0
Combined Terms of Rash (Skin and subcutaneous tissue disorders) | 5 | 4 | 43 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 2 | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 3 | 0 | 0
Tachycardia (Cardiac disorders) | 3 | 0 | 2 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 2 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 7 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 4 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 6 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 15 | 33 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 3 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 1 | 3 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3 | 6 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 10 | 8 | 7 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 9 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 6 | 4 | 0 | 1
Asthenia (General disorders) | 1 | 2 | 2 | 0 | 0
Catheter site haematoma (General disorders) | 1 | 0 | 0 | 0 | 0
Catheter site inflammation (General disorders) | 1 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 2 | 2 | 0 | 0
Chest pain (General disorders) | 0 | 2 | 4 | 0 | 0
Chills (General disorders) | 0 | 2 | 2 | 0 | 0
Fatigue (General disorders) | 6 | 9 | 12 | 0 | 1
Malaise (General disorders) | 0 | 3 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 5 | 0 | 0
Oedema peripheral (General disorders) | 2 | 4 | 5 | 0 | 1
Pain (General disorders) | 0 | 0 | 3 | 0 | 0
Pyrexia (General disorders) | 0 | 3 | 2 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 3 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 3 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 3 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 10 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 3 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 8 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 4 | 6 | 0 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 4 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 5 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 5 | 0 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 2 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 7 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 2 | 0 | 0 | 0
Weight decreased (Investigations) | 3 | 5 | 4 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 2 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 5 | 9 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 3 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 15 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 7 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 5 | 3 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 5 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 6 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 2 | 9 | 0 | 0
Headache (Nervous system disorders) | 2 | 5 | 3 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 3 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 4 | 7 | 0 | 0
Depression (Psychiatric disorders) | 1 | 6 | 4 | 0 | 0
Insomnia (Psychiatric disorders) | 5 | 3 | 7 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 13 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 7 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 6 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 8 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 18 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 9 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 6 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 3 | 26 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All parties agree to submit all manuscripts or abstracts to all other parties 30 days prior to submission. This will enable all parties to protect proprietary information and to provide comments based on information that may not yet be available to other parties. The sponsor may request a delay in publication if there are important intellectual property concerns relating to publication, but does not have the right to suppress publication of the study results indefinitely.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT02186301/Prot_SAP_000.pdf